CLINICAL TRIAL: NCT04763967
Title: A Multi-center, Study of the Non-inferiority of PedSCath Pediatric Sampling Catheter Versus a Retrospective Control Cohort Using Current Standard of Care.
Brief Title: A Study of the PedSCath Pediatric Sampling Catheter Versus Current Standard of Care.
Status: Terminated | Type: Observational
Why Stopped: Slow Enrollment, Recruiting Difficulties
Sponsor: Big Blue Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BBBInc: 0619
Record Dates: First submitted 2020-12-02; First posted 2021-02-21 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Urinary Tract Infections in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Urine samples are collected for both Urinalysis and Urine Culture. Both Urinalysis samples and Urine Culture are retained for 1 Week.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- PedSCath: Subjects in this arm will be catheterized with the PedSCath Pediatric Urinary Cather.
  Interventions: Device: PedSCath Pediatric Urinary Catheter
- Retrospective Control: Generated from 2016 and 2018 anonymized subject data from the clinical sites.
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: PedSCath Pediatric Urinary Catheter — PedSCath Pediatric Sampling Catheter is a pediatric sampling catheter. The product is supplied as a catheter and syringe. PedSCath Pediatric Sampling Catheter is manufactured by Medical Murray Inc. for Big Blue Biotech. The device consists of a blend of LDPE/Elvax/Crodamide.
  Other Names: Wiygul Catheter
  Groups: PedSCath
Device: Standard of Care — Current Standard of Care for pediatric patients
  Groups: Retrospective Control

SUMMARY:
This is a retrospectively-controlled clinical trial that will examine the rate of positive UTI cases among pediatrics entered into the Emergency Department and whose urine is withdrawn using the PedSCath Pediatric Sampling Catheter. The rate of postive UTI will be compared against the control population, whose urine withdrawal would have been performed with Standard of Care devices.

DETAILED DESCRIPTION:
This will be a multi-center, retrospective-controlled, clinical trial.

Anonymized retrospective data from two clinical sites, NewYork-Presbyterian Queens and Weill Cornell Medical College, from 2016 and 2018 will be used to define the control subject population, who were assessed for urinary tract infection (UTI) based on a urine sample taken according to Standard of Care (SoC).

Subjects entering the emergency department (ED) generally require that a urine specimen is obtained and tested to determine whether there is an active infection in the bladder. Emergency department personnel will confirm the possibility of UTI based on symptoms and inform the parents/guardians of the potential for study participation using the PedSCath. The physician will assess the subject based on Inclusion and Exclusion criteria, including non-toilet training and an upper age limit of 3 years. If determined that the subject meets inclusion/exclusion criteria, the physician will inform the parents/guardians of the subject about the study and request informed consent if the parents/guardians wish their child to participate.

Following the granting of Informed Consent, subjects will be enrolled in the study within the treatment arm and a urine sample of 2-3 ml will be taken via the PedSCath. All study assessments, from enrollment through urine sample collection, will occur over a single visit to the ED. Per standard of care, any treatment following the diagnosis will be performed by hospital staff based on physician assessment. Up to 3 run-in subjects per PedSCath user will be treated with PedSCath to allow PedSCath users to become familiar with PedSCath mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 3 years of age or younger.
* Subject is non-toilet trained, as communicated by subject's parent/guardian.
* Subject is presenting to the emergency department with symptoms for UTI, as described by AAP guidelines (Newborns with UTI may present with jaundice, sepsis, failure to thrive, vomiting, or fever. In infants and young children, typical signs and symptoms include fever, strong-smelling urine, hematuria, abdominal or flank pain, and new-onset urinary incontinence) or as determined by PI.
* Subject's parent/guardian is able to provide informed consent.

Exclusion Criteria:

* Any subject with known underlying abnormalities to the genitourinary tract (e.g. prenatal hydronephrosis).
* Any subject who has had prior genitourinary tract or abdominal surgery.
* Any subject who is toilet trained (i.e. able to provide a clean catch urine sample).
* Any subject with an active rash or skin lesion in the suprapubic area.
* Any subject with a known allergy to LDPE, Elvax, or Crodamide plastics.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prospective cohort subjects will enter the emergency department presenting symptoms of UTI. The Control group will be retrospectively enrolled by gathering data through anonymized 2016 and 2018 subject data gathered from the study's clinical sites.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness endpoint is the proportion of PedSCath subjects with positive UTI diagnosis versus that of Control subjects. | Through study completion, an estimation of 1 year.
  The primary effectiveness endpoint is the proportion of PedSCath subjects with positive UTI diagnosis versus that of Control subjects. The objective is to demonstrate a lower rate of positive urinalysis/urine culture results in the PedSCath cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Evan M Haynes, MA, Study Chair — Big Blue Biotech, Inc.
Locations (1):
- NewYork-Presbyterian Queens, New York, New York, United States